CLINICAL TRIAL: NCT01705158
Title: Phase Ib / II Trial Evaluating the Association Myocet ® - Carboplatine in Patients Having a Cancer of the Ovary in Relapse, Sensitive to the Platinum
Brief Title: Myocet ® - Carboplatine in Ovarian Cancer in Relapse, Sensitive to the Platinum
Acronym: MYCA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYCA (GINECO-OV220); 2012-001999-10 (EudraCT Number)
Record Dates: First submitted 2012-10-01; First posted 2012-10-12 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer in relapse; sensitive in platin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carboplatin and liposomal doxorubicin (Experimental): carboplatin and liposomal doxorubicin in ovarian cancer in realapse
  Interventions: Drug: carboplatin and liposomal doxorubicin

INTERVENTIONS:
Drug: carboplatin and liposomal doxorubicin — Carboplatin AUC5 and liposomal doxorubicin 40 or 50 mg/m2, IV (in the vein) on day 1 of each 28 day cycle. Number of Cycles: 6 or until progression or unacceptable toxicity develops.
  Other Names: carboplatin; liposomal doxorubicin, Myocet

SUMMARY:
The purpose of this study is to determine the efficacy and the safety of the association of carboplatine and liposomal doxorubicin in patient with ovarian cancer in relapse, sensitive to platin.

DETAILED DESCRIPTION:
In front of a shortage of Caelyx, the implementation of an alternative treatment must be considered to treat patients with ovarian cancer in relapse, sensitive to platin: associate the carboplatin with another drug of the family of the doxorubicin: liposomal doxorubicin (Myocet®).

ELIGIBILITY:
Inclusion Criteria:

* First or second relapse of a carcinoma of the ovary, the fallopian tubes or the peritoneal tissue histological proved.
* Interval without progress > 6 months after the last administration of a salt of platinum(deck).
* Measurable Disease (according to the criteria RECIST 1.1) or an assessable disease according to CA-125 (according to the criteria of the GCIG).
* Satisfactory biological Balance sheet(Assessment), according to the following criteria:

  * Neutrophiles > 1,5x 109/L, Plaques > 100 x 109/L, Haemoglobin > 9,0 g/dL.
  * Bilirubine < 1.5 x LSN (Normal Superior Limit), transaminases and alkaline phosphatase < 2. 5 x LSN.
  * Creatinin clearance > 50 mL/min calculated according to the formula of Cockroft-Gault or MDRD.
* Performance status < 2.
* Life expectancy of at least 12 weeks.
* Age > 18 years.
* Capacity to follow the protocol.
* Consent signed before any procedure of inclusion.
* Membership in a national insurance scheme.

Exclusion Criteria:

* Tumor of mild histology or borderline, or malignant not epithelial tumor of the ovary, the fallopian tubes or the peritoneal tissue(eg. tumor of germ cells, tumor of the sexual cords and the stroma).
* History of abdominal or pelvic radiotherapy.
* Patient having received more than 2 lines of chemotherapy.
* Patient in 3rd relapse or more.
* History of another malignant tumor during the last 5 years, with the exception of a carcinoma in situ by the neck of the womb or by a squamous-cell carcinoma of the skin treated in a adequate way or any solid tumor considered in forgiveness completes without relapse for at least 5 years.
* Patients having a stubborn illness in the platinum, (eg. progress during the last chemotherapy or in 6 months following the last administration of platinum).
* Occlusive or sub-occlusive disease or presence of symptomatic intellectual metastases.
* Heart disorder dissuading the use of an anthracycline.
* Left venticular ejection fraction (LVEF) defined by MUGA/ECHO < 50%.
* Wait presenting a severe infection.
* Woman old enough to procreate not using adequate contraceptive method.
* Concomitant disease not allowing a surgery and/or a chemotherapy.
* Pathology severe or concomitant not compatible with the taking of the study treatment or the participation of the patient in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Determine the control disease rate in 1 year | 12 months
  To determine the proportion of not progressive patients in 1 year (rate of control of the disease or the rate of not progress in 12 months)

SECONDARY OUTCOMES:
To estimate the rate of objective answer (CR/PR) | 2,5 years
  * To estimate the survival without progress (PFS)
  * To estimate the overal survival (OS)
  * To estimate the profile of toxicity of the association.
  * Quality of life.
  * Validation of the clearance of CA-125 as predictive marker of the efficiency of the treatment and as factor forecast of the survival.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles FREYER, Dr, Principal Investigator — Hospices Civiles de Lyon
Locations (42):
- France (42):
  - Centre de Radiothérapie et d'Oncologie, Agen
  - Centre Paul Papin, Angers
  - Hôpital jean Minjoz, Besançon
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Hôpital Morvan - Centre Hospitalier Universitaire, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Hôpital André Mignot, Le Chesnay
  - Centre Hospitalier du Mans, Le Mans
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Hopital de Scorff, Lorient
  - Centre Léon bérard, Lyon
  - Hopital privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Catherine de Sienne, Nantes
  - Polyclinique KENVAL - Site de Valdegour, Nîmes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Groupe Hospitalier Saint-Joseph, Paris
  - Hopital des Diaconesses, Paris
  - Centre Hospitalier Général de Pau, PAU Universite
  - Clinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - Centre intercommunal de Quimper, Quimper
  - Institut Jean Godinot, Reims
  - Clinique Armoricaine, Saint-Brieuc
  - Centre hospitalier privé de Saint Grégoire, Saint-Grégoire
  - ICO René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Institut cancérologuie de la loire, Saint-Priest-en-Jarez
  - Centre de Radiothérapie - Clinique Sainte-Anne, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier General de Valenciennes, Valenciennes
  - Centre d'oncologie Saint-Yves, Vannes
  - Centre Hospitalier Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Romeo C, Joly F, Ray-Coquard I, El Kouri C, Mercier-Blas A, Berton-Rigaud D, Kalbacher E, Cojocarasu O, Fabbro M, Cretin J, Zannetti A, Abadie-Lacourtoisie S, Mollon D, Hardy-Bessard AC, Provansal M, Blot E, Delbaldo C, Lesoin A, Freyer G, You B. Non-pegylated liposomal doxorubicin (NPLD, Myocet(R)) + carboplatin in patients with platinum sensitive ovarian cancers: A ARCAGY-GINECO phase IB-II trial. Gynecol Oncol. 2019 Jan;152(1):68-75. doi: 10.1016/j.ygyno.2018.10.043. Epub 2018 Nov 14. PMID 30446275